CLINICAL TRIAL: NCT01885338
Title: Dietary Supplement N-acetylcysteine (NAC) as a Novel Complementary Medicine to Improve Cognitive Disfunction in Schizophrenia
Brief Title: N-acetylcysteine (NAC) for Improving Cognitive Dysfunction in Schizophrenia
Acronym: NACSZ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: VISN 22 Mental Illness Research, Education, and Clinical Center (U.S. Federal Agency); American Psychiatric Foundation (Unknown)
Responsible Party: Principal Investigator, Michael C. Davis, M.D., Ph.D., Fellow / Physician, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCC 2013-020208
Record Dates: First submitted 2013-06-17; First posted 2013-06-24 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognition; Neurocognition; N-Acetylcysteine; NAC; EEG
MeSH Terms: conditions — Schizophrenia | interventions — Acetylcysteine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetylcysteine (NAC) (Experimental): Capsules containing N-acetylcysteine 600mg, with inactive ingredients of cellulose, L-leucine, and silica used as filler. Dosage is 2 capsules by mouth twice daily for 8 weeks.
  Interventions: Drug: N-acetylcysteine (NAC)
- Inactive placebo capsule (Placebo Comparator): A placebo capsule is used that is identical to the active treatment but lacks NAC. The inactive ingredients in the placebo capsule are cellulose, L-leucine, and silica. Dose is 2 capsules by mouth twice daily for 8 weeks.
  Interventions: Drug: Inactive placebo capsule

INTERVENTIONS:
Drug: N-acetylcysteine (NAC)
  Other Names: N-acetyl-L-cysteine; NAC
  Arms: N-acetylcysteine (NAC)
Drug: Inactive placebo capsule
  Other Names: Placebo capsule; Sugar pill
  Arms: Inactive placebo capsule

SUMMARY:
This study will evaluate the effect of the dietary supplement N-acetylcysteine (NAC) on electrophysiologic (EEG) markers related to cognition, as well as performance on psychological tests measuring cognition. The primary hypothesis is that participants treated with NAC will show improvements in cognitive function, as measured by EEG and performance-based tests.

DETAILED DESCRIPTION:
Schizophrenia is a serious mental illness associated with substantial social and occupational dysfunction. While positive psychotic symptoms of schizophrenia often respond to antipsychotic medications, negative symptoms and cognitive impairment are difficult to treat, necessitating novel interventions. Cognitive deficits are an important treatment target because the degree of cognitive impairment is a critical predictor of work, education, and social functioning.

Glutamatergic receptors are among the most promising biological targets for cognitive-enhancing drugs in schizophrenia. Abnormal glutamatergic signaling has long been thought to be important in the pathophysiology of schizophrenia; specifically, reduced NMDA glutamatergic receptor activity on thalamic inhibitory neurons disinhibits glutamatergic neurons projecting to the cortex, which can cause secondary dopaminergic abnormalities and lead to characteristic symptoms, including cognitive deficits. Many electrophysiological (EEG) biomarkers related to cognitive dysfunction in schizophrenia are thought to be linked to deficient NMDA glutamatergic neurotransmission. Additionally, neuroplasticity is thought to involve glutamatergic signaling. This pattern of linkages suggests that correcting impaired NMDA glutamatergic transmission in schizophrenia could lead to enhanced cognitive function and learning.

In this pilot study, we will focus on a promising dietary supplement approach to address glutamatergic deficits, evaluating its effects by EEG biomarkers and performance-based neurocognitive assessments. N-acetylcysteine (NAC) is a modified amino acid that is commonly used as a dietary supplement because of its antioxidant properties. NAC modulates glutamatergic signaling as follows: In the CNS, glial cells take up NAC via cystine-glutamate antiporters, which in turn leads to increased glutamate efflux into the extracellular space. Extracellular glutamate binds to non-synaptic glutamate receptors such as the metabotropic glutamate receptors (mGluR) type 2/3 and type 5. The net result of these events is a normalization of pathologically elevated cortical glutamate levels.

We will assess EEG biomarkers associated with cognitive deficits in schizophrenia, including a recently-described biomarker for visual cortical plasticity. We will also perform a comprehensive assessment of neurocognition with the MATRICS battery, which could suggest whether certain cognitive domains are sensitive to improvement with NAC therapy.

Our primary aim is to determine whether NAC administration will improve NMDA-dependent EEG abnormalities in schizophrenia. We have 3 hypotheses: (1) NAC administration will increase mismatch negativity amplitude as compared to placebo; (2) NAC administration will increase P300 amplitude as compared to placebo; and (3) NAC administration will increase gamma oscillation power and phase synchronization as compared to placebo. We also will examine whether NAC will improve measures of visual neuroplasticity, performance-based measures of neurocognition, and clinical symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV-TR criteria for schizophrenia.
2. At least 3 months since any psychiatric hospitalization
3. At least 1 month since meeting criteria for having a major depressive episode
4. At least 6 months since any behaviors suggesting any potential danger to self or others
5. Currently prescribed an antipsychotic medication, with dose not varying >50% over 3 months prior to study participation
6. No acute medical problems that could interfere with study participation
7. Chronic medical problems consistently treated and stable for at least 3 months prior to participation
8. Ability to provide informed consent and cooperate with study procedures

Exclusion Criteria:

1. Documented history of IQ less than 70 or severe learning disability
2. History of treatment with electroconvulsive therapy within 6 months prior to study participation
3. History of neurological or neuropsychiatric condition (e.g., stroke, severe traumatic brain injury, epilepsy, etc.) that could confound assessments
4. Documented history of persistent substance abuse or dependence within 3 months prior to study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
EEG: Change in Mismatch Negativity Amplitude | Change from baseline to 8 weeks
  A passive attention auditory oddball paradigm will be used to assess MMN.
EEG: Change in P300 Amplitude | Change from baseline to 8 weeks
  P300 will be measured using an active attention auditory oddball paradigm.
EEG: Change in Gamma Synchrony Evoked Power and Phase Synchronization | Change from baseline to 8 weeks
  Stimuli will consist of 1-msec 93-dB clicks presented in 500-msec trains presented at 40 Hz, in 3 separate blocks with 200 trials per block. Continuous data will be epoched at -100 to 700 ms relative to stimulus onset and baseline corrected to the average of the prestimulus interval. For evoked gamma power analyses, averages will be computed on a minimum of 120 artifact-free epochs in each block. The averaged epochs across the click trains (0-512 msec) will be transformed into power spectra by fast Fourier transform (FFT). The 40-Hz power spectra will be averaged across 36-45 Hz. Time/frequency intertrial coherence analyses will be performed to assess intertrial coherence of the stimulus-driven EEG signals. In this analysis, coherence ranges from 0 (non-phase-locked random activity) to 1 (activity that is fully locked in phase across individual trials). Responses at electrode Fz will be analyzed.

SECONDARY OUTCOMES:
EEG: Change in Visual Cortical Plasticity | Change from baseline to 8 weeks
  The paradigm involves assessing visual evoked potentials (VEPs) before and after exposure to tetanizing visual high-frequency stimulation (HFS).
Change in MATRICS Consensus Cognitive Battery composite score | Change from baseline to 8 weeks
  The MCCB was developed as a standardized method to assess cognition in clinical trials of potential cognitive-enhancing drugs. It consists of ten tests which assess seven cognitive domains (processing speed, attention, working memory, verbal learning, visual learning, problem solving and reasoning, and social cognition).
Change in Positive and Negative Syndrome Scale (PANSS) total score | Change from baseline to 8 weeks
  This is a widely-used instrument that assesses 30 different symptoms (categorized into positive, negative, and general psychopathology) on a scale from 1 to 7, based on clinical interview.
Change in Clinical Assessment Interview for Negative Symptoms (CAINS) scores | Change from baseline to 8 weeks
  The CAINS is comprised of two subscales that assess the major negative symptom subdomains: 1) Motivation and Pleasure and 2) Expression. This instrument is administered in a semi-structured clinical interview and each of 13 items is rated on a scale ranging from 0 (no impairment) to 4 (severe deficit).

OTHER OUTCOMES:
MIRECC Global Assessment of Functioning (MIRECC GAF) | 4 weeks, 8 weeks
  This is a version of the Global Assessment of Functioning scale in which occupational functioning, social functioning, and symptom severity are scored on a scale of 1-100, with lower scores indicating more impairment in each of the three domains.
Clinical Global Impression (CGI-S and CGI-I | 4 weeks, 8 weeks
  The CGI-S (severity scale) is a widely-used rating scale in which the clinician rates the severity of the subject's mental illness, relative to their past experience with patients with the same diagnosis, on a scale from 1-7, with 1 = normal, not at all ill and 7 = extremely ill. The CGI-I (improvement scale) requires the clinician to rate on a scale from 1-7 how much the mental illness has improved or worsened, relative to a baseline state at the beginning of the intervention, where 1 = very much improved and 7 = very much worse.
Udvalg for Kliniske Undersøgelser (UKU) Side Effects Rating Scale: | 2 weeks, 4 weeks, 8 weeks
  This scale was developed as a comprehensive side effect rating scale for psychopharmacologic medications, with 48 side effects organized into categories.
Barnes Akathisia Scale (BAS) | 4 weeks, 8 weeks
  The most widely-used rating scale to assess the presence and severity of akathisia, the BAS comprises 4 items that rate objective and subjective awareness, subjective distress, and global clinical assessment of akathisia.
Columbia-Suicide Severity Rating Scale (C-SSRS) | 2 weeks, 4 weeks, 8 weeks
  This scale was developed as a screening tool to assess ideation and behaviors associated with suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Marder, M.D., Principal Investigator — VA Greater Los Angeles; Michael C Davis, M.D., Ph.D., Principal Investigator — VA Greater Los Angeles
Locations (1):
- VA West Los Angeles Healthcare Center, Los Angeles, California, United States

REFERENCES:
- [Background] Berk M, Malhi GS, Gray LJ, Dean OM. The promise of N-acetylcysteine in neuropsychiatry. Trends Pharmacol Sci. 2013 Mar;34(3):167-77. doi: 10.1016/j.tips.2013.01.001. Epub 2013 Jan 29. PMID 23369637
- [Background] Cabungcal JH, Steullet P, Kraftsik R, Cuenod M, Do KQ. Early-life insults impair parvalbumin interneurons via oxidative stress: reversal by N-acetylcysteine. Biol Psychiatry. 2013 Mar 15;73(6):574-82. doi: 10.1016/j.biopsych.2012.09.020. Epub 2012 Nov 7. PMID 23140664
- [Background] Shungu DC. N-acetylcysteine for the treatment of glutathione deficiency and oxidative stress in schizophrenia. Biol Psychiatry. 2012 Jun 1;71(11):937-8. doi: 10.1016/j.biopsych.2012.03.025. No abstract available. PMID 22579304
- [Background] Carmeli C, Knyazeva MG, Cuenod M, Do KQ. Glutathione precursor N-acetyl-cysteine modulates EEG synchronization in schizophrenia patients: a double-blind, randomized, placebo-controlled trial. PLoS One. 2012;7(2):e29341. doi: 10.1371/journal.pone.0029341. Epub 2012 Feb 22. PMID 22383949
- [Background] das Neves Duarte JM, Kulak A, Gholam-Razaee MM, Cuenod M, Gruetter R, Do KQ. N-acetylcysteine normalizes neurochemical changes in the glutathione-deficient schizophrenia mouse model during development. Biol Psychiatry. 2012 Jun 1;71(11):1006-14. doi: 10.1016/j.biopsych.2011.07.035. Epub 2011 Sep 25. PMID 21945305
- [Background] Dean O, Giorlando F, Berk M. N-acetylcysteine in psychiatry: current therapeutic evidence and potential mechanisms of action. J Psychiatry Neurosci. 2011 Mar;36(2):78-86. doi: 10.1503/jpn.100057. PMID 21118657
- [Background] Berk M, Copolov D, Dean O, Lu K, Jeavons S, Schapkaitz I, Anderson-Hunt M, Judd F, Katz F, Katz P, Ording-Jespersen S, Little J, Conus P, Cuenod M, Do KQ, Bush AI. N-acetyl cysteine as a glutathione precursor for schizophrenia--a double-blind, randomized, placebo-controlled trial. Biol Psychiatry. 2008 Sep 1;64(5):361-8. doi: 10.1016/j.biopsych.2008.03.004. Epub 2008 Apr 23. PMID 18436195